CLINICAL TRIAL: NCT01518205
Title: HELP-Apheresis in Diabetic Ischemic Foot Treatment (H.A.D.I.F): a RCTrial to Evaluate the Effect of LDL-apheresis on the Recovery of Diabetic Ulcers in Patients With Peripheral Vasculopathy Not Susceptible to Revascularization.
Brief Title: HELP-Apheresis in Diabetic Ischemic Foot Treatment (H.A.D.I.F)
Acronym: HADIF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universita di Verona (Other)
Responsible Party: Principal Investigator, Maria Grazia Zenti, Maria Grazia Zenti,MD, Division of Endocrinology and Metabolic Diseases, University Hospital of Verona, Universita di Verona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MZenti HADIF
Record Dates: First submitted 2012-01-22; First posted 2012-01-25 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2017-01

CONDITIONS: Foot Ulcers; Arteriosclerosis Obliterans; Diabetes Mellitus
Keywords: diabetic foot ulcers,; peripheral arterial disease,; heparin-induced extracorporal lipid apheresis.; inflammatory markers; type 2 diabetes; LDL-cholesterol
MeSH Terms: conditions — Foot Ulcer; Arteriosclerosis Obliterans; Diabetes Mellitus; Diabetic Foot; Peripheral Arterial Disease; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- LDL-apheresis and TT (Experimental): The patient of the experimental Arm, in addition to Traditional Therapy (TT), will undergo a cycle of 10 LDL-apheresis session.
  Apheretic treatment scheme: 10 apheretic session carried out as follow: first and second apheresis with a 3 days interval (i.e. 2 treatment in one week), then one session per week (every 7 days).
  To perform the treatment, the forearm surface veins will be punctured by means of 17 Ga needles, as an alternative a two-ways CVC will be used.
  Interventions: Device: LDL-apheresis
- Traditional Treatment (No Intervention): All patients will receive the traditional treatment for the ulcer healing Standardized medication.
  All lesions taken into consideration will be treated in a standardized way, with a different approach according to the presence of a possible infection.
  The evolution of lesions might be documented by means of mapping the same by drawing their profiles on an Opsite film.
  antibiotics therapy (according to antibiogram). Anti-platelet therapy. Statin therapy.

INTERVENTIONS:
Device: LDL-apheresis — The patient of the Arm "LDL-apheresis" in addition to standard therapy, will undergo a cycle of LDL-apheresis.
  LDL-apheresis will be performed with B.Braun Avitum H.E.L.P. System. Apheretic treatment scheme: 10 apheretic sessions carried out as follows: the first 2 with a 3 day distance (i.e. 2 treatments in one week), successively 1 session per week (every 7 days).
  To perform the treatment, the forearm surface veins will be punctured by means of 17 Ga needles, as an alternative a two-ways CVC will be used.
  Other Names: H.E.L.P. apheresis; TT: traditional therapy
  Arms: LDL-apheresis and TT

SUMMARY:
Diabetic foot (DF) is a common, severe and costly complication of diabetes. DF is underlied by neuropathy, atherosclerosis of distal arteries and infection, which result in tissue ulcers and necrosis. Alterations in microcirculatory function and in blood rheology may concur in causing tissue damage.

In recent years there has been accumulating evidence that LDL apheresis (LA) does not only reduce cholesterol but also has a series of pleiotropic effects that improve the microcirculation, increasing peripheral tissue perfusion.

HADIF is a randomized, multicentric, prospective clinical study aimed at assessing the effect of LDL apheresis treatment in association with traditional therapy for ulcers, in patients with an ischemic diabetic foot ulcer (class I and II Texas Wound Classification System)and peripheral vasculopathy not susceptible to revascularization. A total of 132 patients will be enrolled. Participants will be centrally randomized to receive traditional therapy alone (TT) or in association with LA. TT includes standard medication of ulcers, antiaggregant therapy and statins. LA will be performed with HELP system, for a total of 10 sessions in 9 weeks. The primary end-point of the study is ulcer healing; secondary endpoints include improvements of peripheral oxygenation, resolution of pain, reduction of circulating inflammatory markers, cardiovascular events during one year's follow-up.

This clinical Study has been approved by local EC on 25 may 2011 (Study number 1953).

TO BE NOTED: since diabetic patients in our "Diabetic-Foot UNIT" often presented foot ulcers more severe than class II Texas, a formal amendment has been submitted to EC for recruiting patients with diabetic foot ulcer of class III Texas. The amendment was already approved on 5 may 2012.

DETAILED DESCRIPTION:
Aim of the protocol is to evaluate the effect of LDL-apheresis in combination with traditional therapy, on the recovery of diabetic ulcers in patients suffering from diabetic ischemic foot and peripheral vasculopathy that cannot be revascularized.

Patients who qualify for the study will be randomized to the traditional treatment combined to apheresis (Experimental Arm) or to the standard treatment only (control Arm).

The randomization stratified according to the lesion gravity level (class TEXAS I vs II vs III),allocation 1:1. The randomization list will be generated by the statistic software "Stata 11". The lists of randomization (one list for each class TEXAS ) will be generated and will be stored by the coordinator centre. When a patient satisfies the study inclusion criteria, will be contacted the coordinator centre (by phone/mail) for group allocation.

132 patients will be enrolled (66 patients in experimental arm, 66 patients in control arm).

Traditional Therapy (TT) includes standard medication of ulcers, antiaggregant therapy and statins.

LDL-apheresis (intervention Arm) will be performed with HELP system, for 10 session in 9 weeks.

Blood samples will be collected (at basal, and after 3-6-9-12 months) in order to determine the following parameters: glycaemia, insulin, glycated haemoglobin, microalbuminuria/creatinuria,CBC, fibrinogen, total cholesterol, HDL-cholesterol, LDL-cholesterol, Triglycerides, Lp(a), C-reactive protein (CRP), pentraxin3 (PTX3).

Furthermore, in patients of experimental arm, blood samples will be collected at basal and at the end of LDL-apheresis sessions no. 2 and 10 in order to determine CBC, fibrinogen, total cholesterol, HDL-cholesterol, LDL-cholesterol, Triglycerides, Lp(a), CRP, PTX3 (time schedule, after 1 and 9 weeks).

The value of the lab tests obtained at the end of apheresis will be normalized due to a possible hemodilution, according to the following formula:

F dil= (1 - Htc pre-apheresis) / ( 1 - Htc post-apheresis). Xcorrect = Xmeasured * Fdil.

Ulcer evaluation: staging according to Texas Wound classification System and ulcer surface evaluation (diameter, mapping of the lesions by means of drawing their profiles on Opsite film; digital picture): at basal, at 9th week and after a 3-6-9-12 month follow-up.

The ulcers evolution will be "in blind" monitored by an evaluator who will check ulcer-map and digital picture without knowing to which randomization arm they belong.

Transcutaneous oximetry: basal, at 4th week (i.e. after the 5th apheretic session). at 9th week (at the end of the 10 apheresis sessions) and after the next 3-6-9-12 month follow-up.

Questionnaire on quality of life (SF36): basal, at 9th week (at the end of the 10 apheresis sessions) and after the next 6-12 month follow-up.

Pain intensity rate (verbal numeric range) basal, at 9th week (at the end of the 10 apheresis sessions) and after the next 3-6-9-12 month follow-up.

Doppler flowmeter : basal, at 9th week (at the end of the 10 apheresis sessions) and in the subsequent follow-up at 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic patients
* Ischemic diabetic ulcers (class I, II and III Texas Wound Classification System);
* documented peripheral vasculopathy with at least a previous event of failed revascularization (no ulcer healing).

Exclusion Criteria:

* Patient refusal to participate
* BMI > 35 kg/m2
* Ischemic diabetic ulcers class III Texas Wound Classification System
* Patients presenting a bleeding diathesis, malignant tumor, heart failure not allowing extracorporeal technique.
* Haemodialysis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2012-02; Primary Completion 2015-09 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects obtaining the ulcer healing (Class 0A according to TEXAS classification) after 12 month from the study starts. | 12 months
  Ulcer evaluation: staging according to Texas Wound classification System and ulcer evaluation (surface diameter, mapping of the lesions by means of drawing their profiles on Opsite film,and digital picture), at basal, at 9th week and after a 3-6-9-12 month follow-up.

SECONDARY OUTCOMES:
Improvement of the peripheral oxygenation evaluated by means of transcutaneous oximetry measurement at foot level: TcP O2 (mmHg). | basal, at 4th and 9th week and after 3-6-9-12 month follow-up
Evaluation of pain level variation (verbal numeric range; score from 1 to 10) | basal, at 4th and 9th week and after 3-6-9-12 month follow-up
Lowering of circulating inflammation markers (C Reactive Protein, Fibrinogen). CRP plasmatic concentration (mg/L) and fibrinogen (g/L) | at the beginning of the study and respectively after 3 - 6 - 9 e 12 months.
Rate of cardiovascular events in the observation period (1-year follow-up). | 12 months
proportion of subjects with minor amputation (only toe or part of the foot removed)- in agreement with the approved amendment | 12 months
proportion of subjects with major amputation (these are usually below the knee or above the knee)- in agreement with the approved amendment | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Maria Grazia Zenti, MD, Principal Investigator — Division of Endocrinology and Metabolic Diseases, University Hospital of Verona; Enzo Bonora, MD, PhD, Study Director — Division of Endocrinology and Metabolic Diseases, University Hospital of Verona
Locations (1):
- universita Verona, Verona, Verona, Italy

IPD SHARING:
Plan to Share IPD: No